CLINICAL TRIAL: NCT03879564
Title: Efficacy of Ketamine-fentanyl VS Fentanyl for Analgosedation in Postoperative Ventilated SICU Patients
Brief Title: Ketamine-fentanyl VS Fentanyl for Analgosedation in SICU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Karuna Wongtangman, principle investigator, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Si783/2018
Record Dates: First submitted 2019-03-11; First posted 2019-03-18 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Critically Ill; Pain, Postoperative
MeSH Terms: conditions — Critical Illness; Pain, Postoperative | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: ketamine and normal saline will be filled in 50-ml syringe and will be administered in the same condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Placebo Comparator): 0.9% NaCl IV bolus 0.3 ml/kg then drip 0.09 ml/kg/hr
  Interventions: Drug: Normal saline
- ketamine (Experimental): ketamine in NSS (1 mg/ml) IV bolus 0.3 ml/kg then drip 0.09 ml/kg/hr
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — ketamine in NSS (1 mg/ml) IV bolus 0.3 ml/kg then drip 0.09 ml/kg/hr
  Arms: ketamine
Drug: Normal saline — NSS IV bolus 0.3 ml/kg then drip 0.09 ml/kg/hr
  Arms: control

SUMMARY:
This is a randomized, double-blinded study to evaluate the analgosedative effect of ketamine in a surgical intensive care unit. The patients who will receive continuous fentanyl infusion for either pain control or sedation will be recruited in this trial. Fentanyl will be titrated with initial loading doses of 20 mcg until the numeral rating scale(NRS) less than 4 or critical care pain observation tool (CPOT) less than 3 or Richmond agitation sedation score (RASS) -2-0. Then the patients will be randomised in to receive saline infusion in control group (Group C) or ketamine infusion in ketamine group (Group K). Ketamine will be administered with an initial bolus of 0.3 mg/kg followed by a perfusion of1.5 mcg/kg/min during the first 48 h. The dose of fentanyl will be protocolized adjusted according to NRS or CPOT or RASS. We tested the research hypothesis that low-doseketamine infusion is associated with a reduced fentanyl dose without increased vulnerability to its psychotropic effects.

DETAILED DESCRIPTION:
Upon SICU admission, patient eligibility will be assessed, and informed consent will be obtained. A fentanyl bolus will be titrated by attending physicians to reach the target of patients' NRS pain scores at < 4 (self-report) or CPOT scores < 3 (unable to self-report pain) or patients' Richmond agitation and sedation scale (RASS) scores between -2 and 0.

After enrollment, patients will be randomly assigned in a 1:1 ratio by their sequential number of enrollment to receive either ketamine infusion (Group K) or placebo (Group C) together with fentanyl at 20 mcg/hr, initially. Randomization will be performed using a computer-generated randomization table derived from www.randomization.com. This process will be performed by an investigator (K.W.) who has no other role in patient enrollment or management. The other investigators, the patients, the patients' relatives, the attending physicians, and the nurses will all blinded to the study assignment. The study drug (ketamine or placebo) will be prepared by a pharmacist, who has no other role in the trial. The study drugs are packaged in identically shaped containers labeled with sequential numbers according to the randomization table order. For the study drug, 50 mg of ketamine is mixed with 50 ml of 0.9% NaCl (NSS), giving a final ketamine concentration of 1 mg/ml. For the placebo comparator, 50 ml of NSS will be prepared. The study drug will infuse via either peripheral line or central venous catheter (when available) at an individually adjusted rate according to the patient's body weight to achieve a dose of ketamine of 1.5 mcg/kg/min. The study drug will infuse for a period of 48 hours or until discontinue if narcotic medication without titration in both groups.

All eligible patients will receive narcotic and sedative medication according to the pain and sedation protocol. This included infusion of narcotic medication (fentanyl) and sedative medication to keep target NRS scores at < 4 and RASS scores between 0 and -2. Additional 20-mcg fentanyl IV bolus every 10 minutes will be administrated if needed. If more than 2 boluses are given per hr, the fentanyl rate will be increased by 10 mcg/hr to achieve pain and sedation goals. Blinded nurses will record pain scores, RASS, and medication doses every 4 hours.

Fentanyl IV infusion will be held if the RASS score is less than -2, indicating oversedation. If fentanyl is not administered for over one hour and the patient's RASS score remained below -2, the study drug will be discontinued.

A telephone follow-up will be conducted 12-60 months after ICU discharge using the Thai version of the Posttraumatic Symptom Scale (PTSS-10 questionnaire) to screen for the occurrence of PTSD as well as traumatic memories in the ICU. The interviews will be conducted by a research team unaware of the patients' group assignment.

Primary outcome is fentanyl consumption within 24 hours after randomization. Secondary outcomes are adverse effects of ketamine which will be assessed during study drug administration and long-term follow up (12-60 months) of the patient using questionnaires on traumatic memories from their ICU stay and post-traumatic stress disorder (PTSD) screening questionnaire (PMID: 10470573).

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years.
* Need ICU care
* Need continuous iv fentanyl as an sedative of analgesia drug

Exclusion Criteria:

* Pregnant women
* Known allergy to ketamine
* Severe cardiovascular disorders (ejection fraction< 30%, acute myocardial infarction, decompensated heart failure, significant tachyarrhythmia)
* Acute psychosis
* coma patient
* receive
* Renal insufficiency (creatinine clearance < 30 mL/min)
* Unable to assess pain with either NRS or CPOT
* Neurosurgery/ CVT patients/ trauma patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
fentanyl consumption | 24 hours after initial fentanyl infusion
  the amount of fentanyl in microgram/kg in the patients who receive ketamine compare with who receive NSS

SECONDARY OUTCOMES:
Psychomimetic adverse effects | 72 hours after admitted to ICU
  incidence of delirium assess by CAM ICU hallucination nightmare
Duration of mechanical ventilation | 30 days after admitted to ICU
ICU length of stay | 30 days after admitted to ICU
bowel motility | 72 hours after admitted to ICU
  first pass stool day
cardiovascular effect | 72 hours after admitted to ICU
  Number of participants that experience episode of unexplained hypertension (sustained (> 30 min) increase in MAP + 25% from baseline) during ketamine infusion
cardiovascular effect | 72 hours after admitted to ICU
  Number of participants that experience tachyarrhythmia;- Supraventricular/ventricular tachycardia during ketamine infusion
cardiovascular effect | 72 hours after admitted to ICU
  Number of participants that experience atrial fibrillation with rapid ventricular response, rate > 110 bpm during ketamine infusion
cardiovascular effect | 72 hours after admitted to ICU
  Number of participants that experience sinus tachycardia rate >130 bpm
Long-term effect | 12 to 60 months after ICU discharge
  Number of traumatic memories that might be associated with ketamine per participant: Nightmares, severe anxiety or panic, and feeling of suffocation.
Long-term effect | 12 to 60 months after ICU discharge
  Number of participants that has traumatic memories associated with severe pain.
Long-term effect | 12 to 60 months after ICU discharge
  Number of participants that screening test positive for PTSD

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine Siriraj hospital, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kitisin N, Raykateeraroj N, Hemtanon N, Kamtip P, Thikom N, Azimaraghi O, Piriyapatsom A, Chaiwat O, Eikermann M, Wongtangman K. Effect of Low-Dose Ketamine Infusion in the Intensive Care Unit on Postoperative Opioid Consumption and Traumatic Memories After Hospital Discharge: A Randomized Controlled Trial. Anesth Analg. 2025 Sep 1;141(3):598-607. doi: 10.1213/ANE.0000000000007419. Epub 2025 Feb 5. PMID 39908192